CLINICAL TRIAL: NCT05690763
Title: Quantitative Assessment of the Efficacy of Two Irrigation Activation Systems in Reducing the Bacterial Load in Teeth With Post-treatment Apical Periodontitis: A Clinical Study
Brief Title: Quantitative Assessment of the Efficacy of Two Irrigation Activation Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seyda Ersahan, DDS, PhD (Other)
Responsible Party: Sponsor-Investigator, Seyda Ersahan, DDS, PhD, The Antimicrobial Efficacy of Sweeps Laser Compared to Ultrasonically Activated Irrigation and Needle Irrigation in Posterior Teeth With Apical Periodontitis: A Clinical Study, Istanbul Medipol University Hospital
Organization: Istanbul Medipol University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Microbial analysis
Record Dates: First submitted 2022-12-16; First posted 2023-01-19 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Periapical Periodontitis; Polymerase Chain Reaction; Enterococcus Faecalis Infection; Irrigation Activation
MeSH Terms: conditions — Periapical Periodontitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- XP-endo Finisher (Experimental): use of XP-endo Finisher
  Interventions: Other: XP-endo Finisher to use irrigation activation
- EndoActivator (Experimental): use of EndoActivator
  Interventions: Other: EndoActivator to use irrigation activation

INTERVENTIONS:
Other: XP-endo Finisher to use irrigation activation — XPF : The canals were flushed with 2.5 mL 2.5% NaOCl for 30 s and activated by a XPF instrument that was placed in the canal to 1 mm short of the WL and powered by the motor at 800 rpm (1 N-cm torque) for 30 s according to the manufacturer's instructions. Then the canals were rinsed with 2.5 mL of 2.5% NaOCl, followed by activation of the substance with the XPF instrument for 30 seconds, the same way as above. A new XP-endo Finisher file was used for each canal.
  Arms: XP-endo Finisher
Other: EndoActivator to use irrigation activation — The root canals were irrigated with 2.5 mL of 2.5% NaOCl for 30 s, followed by sonic activation of this solution with EndoActivator red tip size #25/0.04, inserted into the root canal 1 mm short of the WL, at 10,000 cpm/min. for 30 seconds. The EA polymer tip moved vertically from apical to coronal part of the canal during activation.
  Arms: EndoActivator

SUMMARY:
Aim of the present study was to determine the intraradicular microbiota of previously root canal-treated teeth with apical periodontitis using droplet digital polymerase chain reaction (ddPCR) and to investigate the antibacterial effectiveness of different irrigation activation methods [ XP-endo Finisher and EndoActivator ] that will make classical chemomechanical preparation more effective. This superiority, parallel, randomized clinical trial was conducted in the clinic of the Endodontic Department, Faculty of Dentistry, Istanbul Medipol University, Istanbul. 20 patients with posttreatment apical periodontitis (one tooth each) were randomly allocated into two groups according to the used (n=10, for each): the EA group (A) or the XPF group (B). Total bacterial loads, as well as the amount of Enterococcus faecalis (E.faecalis) were determined before (S1) and after (S2) chemomechanical preparation and finally, after intracanal medication (S3) by means of ddPCR.

DETAILED DESCRIPTION:
Eligibility criteria The study population consisted of 20 patients (9 women and 11 men, aged 19-66 years) presenting to the endodontic clinic at Istanbul Medipol University Dental School, for nonsurgical endodontic retreatment of teeth with apical periodontitis lesions. 20 previously root canal-treated teeth exhibiting clinical and radiographic evidence of chronic apical periodontitis lesions were included in this study. Radiographically, the diameter of the periapical radiolucency ranged from 2 to 7 mm. Teeth with post-treatment apical periodontitis had endodontic therapy completed more than 2 years earlier and required retreatment. Termini of the root canal fillings ranged from 0-4 mm short of the radiographic apex, with no overfilling. The teeth had intact coronal restorations, with no obvious exposure of the root-filling material to the oral cavity. Selected teeth had enough crown structure for adequate isolation with a rubber dam and showed an absence of periodontal pockets or attachment level deeper than 4 mm. Exclusion criteria were also applied, as follows: teeth from patients who had received antibiotics within the previous 3 months or who had any general disease, teeth that could not be properly isolated with rubber dam, teeth with absence of coronary sealing, teeth with periodontal pocket depth >4 mm; and teeth with crown/root fracture. Only one tooth was included from each patient.

Root canal treatment procedures and sampling Rubber dam and an aseptic technique were used throughout the endodontic retreatment. After plaque removal and rubber dam isolation, the operative field was cleaned with 3% hydrogen peroxide and disinfected with 2.5% NaOCl solution. Then, all coronal restorations, posts and carious defects were removed and access preparation was completed when the root canal filling was properly exposed. Afterwards, the tooth (including the pulp chamber), clamp, and adjacent rubber dam were once again disinfected with 2.5% NaOCl, followed by inactivation with 10% sodium thiosulfate in order to avoid interference with bacteriological sampling. Sterility control samples (SR1) were taken from the tooth surface with a sterile Omni Swab (Whatman FTA, Sigma-Aldrich) with an ejectable head. Paper points were transferred to cryotubes containing phosphate buffered saline (PBS) solution stored at -20°C. In each case, a single root canal was sampled in order to confine the microbial evaluation to a single ecological environment. In multirooted teeth, the root with the periapical lesion was selected. If there were periapical lesions in all roots, the wider canal was selected. Two of the canals included in this study were from single-rooted teeth, 3 were buccal canals in maxillary premolars, 1 palatal canal in maxillary molar, and 10 distal canals in mandibular molars.

Old root fillings were removed using Gates-Glidden drills (Dentsply Maillefer, Ballaigues, Switzerland) and endodontic files without the use of chemical solvents. The working length (WL) was established 1-mm short of the apical foramen with an apex locator (Raypex6; VDW GmbH, Munich, Germany), and then periapical radiographs were taken to ensure that all filling material was removed. Irrigation with sterile saline solution was performed in order to remove any remaining materials and to moisten the canal prior to sample collection. Next, the canal was left filled with saline, and a small hand instrument was placed at the WL and used to gently file the canal walls. An initial microbiologic sample (S1) was taken from the root canal with sterile paper points consecutively placed at the WL. Three sterile paper points were inserted into the root canal for sampling. Each paper point was left in the canal for about 1 minute. Both the paper points and the endodontic hand instrument, without the handle, were transferred to cryotubes containing 300 μl of PBS solution stored at -20°C. The samples were transferred to genetic analysis laboratory for further analysis in cold chain.

Root canals were prepared by using the Revo S files and irrigated with 2.5% NaOCl. The canals were apically enlarged to size 35 (AS35) at the working length. Between each instrument change, the root canal was irrigated with 5 ml of 2.5% NaOCl solution by using 30-gauge side-vented needle, which was placed 1 to 2 mm short of working length. Hence, a total of 30 mL of the irrigating solution was used. After instrumentation was completed, the smear layer was removed with 2 mL 17% EDTA, which was left in the canal for 3 min, followed by 2.5% NaOCl. The root canal was dried with sterile paper points and flushed with 2 ml of 10% sodium thiosulfate for 1 min to inactivate the NaOCl solution. Next, a sample (S2) was taken from the canals as described for S1. Following this, the NaOCl was agitated/activated as described below.

XPF group: The instrument XP-Endo Finisher (FKG Dentaire, size #25, taper .00) was cooled down (Endo-Frost; Roeko, Langenau, Germany) in order to keep it straight and measure the WL. The canals were flushed with 2.5 mL 2.5% NaOCl for 30 s and activated by a XPF instrument that was placed in the canal to 1 mm short of the WL and powered by the motor at 800 rpm (1 N-cm torque) for 30 s according to the manufacturer's instructions (in slow up-and-down movements at approximately 7-mm amplitude in continuous rotation). Then the canals were rinsed with 2.5 mL of 2.5% NaOCl, followed by activation of the substance with the XPF instrument for 30 seconds, the same way as above. A new XP-endo Finisher file was used for each canal.

EA group: The root canals were irrigated with 2.5 mL of 2.5% NaOCl for 30 s, followed by sonic activation of this solution with EndoActivator red tip size #25/0.04 (EA; Dentsply Tulsa Dental Specialties, Tulsa, OK), inserted into the root canal 1 mm short of the WL, at 10,000 cpm/min. for 30 seconds. The EA polymer tip moved vertically from apical to coronal part of the canal during activation. Then the same procedure was repeated once more (sonic activation of 2.5 mL of 2.5% NaOCl for 30 seconds) so that the total irrigation with NaOCl and irrigation agitation time with the test devices were 1 min. The total volume of NaOCl used per canal in both groups was 35 mL. In both groups, 5 mL of NaOCl was used and activated for one minute.

Finally, the canals in both groups were dried and rinsed with 2 mL 10% sodium thiosulfate for 1 min. The post activation sample (S3) was obtained in the same way as the pre-activation sample was collected and sent for the PCR analysis. Completion of the root canal treatment proceeded with root filling using lateral condensation of gutta-percha. Access cavities were restored with composite resin, and a final radiograph was taken. All the root canal and microbial sampling procedures were performed by a single experienced endodontist. Total bacterial loads, as well as the amount of Enterococcus faecalis were determined before instrumentation, after instrumentation and use of the irrigation activation systems, by means of droplet digital polymerase chain reaction (ddPCR).

Total bacterial loads, as well as the amount of Enterococcus faecalis were determined before instrumentation, after instrumentation and use of the intracanal medicaments, by means of ddPCR.

Genomic DNA isolation and measurement of DNA concentration DNA was extracted using the QIAamp DNA Mini Kit (Qiagen, Germany) following the protocol recommended by the manufacturer. Before DNA isolation, samples (the tubes with paper points) were digested at 50-60°C BY vortexING for 30s in every 10 min in order to ensure disaggregation of all bacteria into the PBS solution. Afterwards, the paper points were aseptically removed from the suspension and, the bacterial suspension was pelleted by centrifugation for 10 min at 5000 g. The pellet was then resuspended in 180 µl buffer ATL supplied by QIAamp DNA Mini Kit (QIAGEN GmbH, Hilden, Germany) and 20 µl proteinase K (20 mg/ml) was added. Samples were incubated for 3 h at 56°C. Subsequently, total bacterial genomic DNA was isolated according to the protocol of the QIAamp DNA Mini Kit. The final volume of DNA solution of each sample was 150 μL and was taken into account during calculation. DNA concentration (absorbance at 260 nm) was determined with a spectrophotometer (Promega Quantifluor).

Amplification of 16S rRNA genes Primers for Universal and Enterococcus 16S rRNA genes were designed in this study. After DNA extraction of samples with QIAamp DNA Mini Kit, 700-800 bp of 16S rRNA sequences were amplified by using universal E8F forward primer (5'-AGAGTTTGATCCTGGCTCAG-3') and universal E1115R reverse primer (5'-AGGGTTGCGCTCGTTG-3') 59. The final volume of PCR reactions for each isolated bacterial strain was adjusted to 25 µl. The amplification reactions of 16S rRNA genes were performed with the following conditions. 1 cycle of predenaturation at 95°C for 3 minutes, 35 cycles of 95°C for 30 seconds, 55°C for 30 seconds, and 72°C for 30 seconds which continue with a final extension step at 72°C for 10 minutes.

The PCR products were analyzed by electrophoresis using 2% agarose gel (containing ethidium bromide) in Tris/BoratE/EDTA (TBE) buffer, with gels being analyzed under ultraviolet light (at 140V for 20 minutes). Their images were visualized under ultraviolet illumination. In addition, the control and optimization of primers to be used for ddPCR was also done in conventional PCR.

Purification and Sequencing of the 16S rRNA Gene After the PCR reactions, the purification of PCR products is done by hydrolyzing the excess primers and nucleotides with ExoSap-IT (Thermo, PN: 78201.1.ML) containing Exonuclease I and Alkaline Phosphatase enzymes. 2 µl of ExoSap-IT was mixed with 5 µl of PCR product for each sample. The ExoSap reaction is performed at 37 °C for 15 minutes (enzyme activation) followed by 15 minutes (inactivation) at 80 °C. Sequencing reactions were performed by using Bigdye™ Terminator v3.1 cycle sequencing kit (Thermo). The reactions were performed according to the kit manual for all isolated strains.

After purification of the products with Exosap, the sequence reaction was performed with BigDye Terminator v3.1 Cycle Sequencing Kit (Thermo) under the following conditions. After the sequence PCR, BigDye products were purified by colon method. Zymo ZR DNA Sequencing Clean-up Kit (Zymo Research, USA) was used for this process. All samples were purified in accordance with the protocol given in the kit and executed on the 3130XL genetic analyzer.

Droplet Digital PCR (ddPCR) Droplet Digital PCR (ddPCR) was performed using primers designed according to the 16S rRNA region specific to the total bacteria and Enterococcus faecalis species, after sequencing, absolute quantitation from the bacterial species found in the paper-point sample. Primer pairs were 16S-F-5'-AGGGAATCTTCSGCAATGGG-3' and 16S-R-5'-ACGCCCAATAAATCCGGACA-'3 for total bacteria and ENT-F-5'-CGCTTCTTTCCTCCCGAGT-3' and ENT-R-5'-GCCATGCGGCATAAACTG-3' primer pairs for Enterococcus Faecalis. In the PCR reaction, amplicons amplified with unmarked primer pairs were analyzed by labeling with Eva-Green dye. For absolute quantitation of Enterococcus and total 16S rRNA, PCR was performed with two primer pairs from the same sample. 20 µL of PCR mix containing 10 µL of 2X ddPCR EvaGreen Supermix (Bio-Rad, cat. no. 1864034), 9 µL of nuclease-free water, 0.25 µL of both forward and reverse primer and 2 ng of DNA from each sample Thermal cycling conditions were: 95◦C for 5 min, then 40 cycles of 95◦C for 30 s and 60◦C for 1 min and two final steps at 4◦C for 5 minutes and 90◦C for 5minutes with a 4◦C infinite hold. After PCR was completed, the sealed plate was transferred into the plate holder of the QX200 Droplet Reader (Bio-Rad, cat. no. 1864003).

ELIGIBILITY:
Inclusion Criteria:

* root canal-treated teeth exhibiting clinical and radiographic evidence of chronic apical periodontitis lesions.
* Teeth with post-treatment apical periodontitis had endodontic therapy completed more than 2 years earlier and required retreatment.
* Radiographically, the diameter of the periapical radiolucency ranged from 2 to 7 mm.
* Termini of the root canal fillings ranged from 0-4 mm short of the radiographic apex, with no overfilling.
* The teeth had intact coronal restorations, with no obvious exposure of the root-filling material to the oral cavity.
* Selected teeth had enough crown structure for adequate isolation with a rubber dam and showed an absence of periodontal pockets or attachment level deeper than 4 mm.

Exclusion Criteria:

* teeth from patients who had received antibiotics within the previous 3 months or who had any general disease, teeth that could not be properly isolated with rubber dam, teeth with absence of coronary sealing, teeth with periodontal pocket depth >4 mm; and teeth with crown/root fracture. Only one tooth was included from each patient.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2022-09-02 (Actual); Study Completion 2022-12-02 (Actual)

PRIMARY OUTCOMES:
the sequence analysis of 16S rRNA genes by the Sanger sequencing | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: SEYDA ERSAHAN, Assoc.Prof., Principal Investigator — IstanbulMedipol University
Locations (1):
- Istanbul Medipol University, Faculty of Dentistry, Istanbul, Esenler, Turkey (Türkiye)